CLINICAL TRIAL: NCT04597424
Title: Combined Prevention of Sexually Transmitted Infections (STIs) in Men Who Have Sex With Men and Using Oral Tenofovir Disoproxil Fumarate/ Emtricitabine (TDF/FTC) for HIV Pre-Exposure Prophylaxis (PrEP)
Acronym: DOXYVAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 174 DOXYVAC
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Unsafe Sex; Risk-Taking
Keywords: STI infection; PREVENTION
MeSH Terms: conditions — Unsafe Sex; Risk-Taking

STUDY DESIGN:
Intervention Model Description: Arm 1 : doxycycline and Bexsero vaccine Arm 2 : doxycycline and no vaccine Arm 3 : No doxycycline and Bexsero vaccine Arm 3 : No doxycycline and No Bexsero vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- doxycycline and Bexsero® vaccine (Experimental): -doxycycline will be taken by participants as PEP (prophylaxy post exposition) and participants will received Meningococcal B vaccine (Bexsero®) at D0 and M2
  Interventions: Drug: Experimental: doxycycline; Biological: Bexsero® vaccine
- doxycycline (Experimental): -doxycycline will be taken by participants as PEP (prophylaxy post exposition)
  Interventions: Drug: Experimental: doxycycline
- Bexsero® vaccine (Experimental): -Meningococcal B vaccine (Bexsero®) at D0 and M2
  Interventions: Biological: Bexsero® vaccine
- No treatment (No Intervention): -no doxycycline and no Bexsero® vaccine

INTERVENTIONS:
Drug: Experimental: doxycycline — 2 tablets of doxycycline 100 mg (monohydrate form) will be taken orally after each risk sexual intercourse, ideally within 24 hours after sex and no more than 72 hours. PEP should not be taken more than 3 times over a 7 days' period.
  If a participant has risk sexual intercourse for several consecutive days, PEP should be taken at least 48 hours apart and no more than 3 times 2 tablets over 7 days. A maximum of 3 intakes of 2 tablets will be allowed over a period of 7 days.
  Arms: doxycycline; doxycycline and Bexsero® vaccine
Biological: Bexsero® vaccine — 1st injection of Bexsero® vaccine at inclusion visit, 2nd injection at week 8.
  Arms: Bexsero® vaccine; doxycycline and Bexsero® vaccine

SUMMARY:
The study ANRS 174 Doxyvac is a clinical trial that will use Combined Prevention of Sexually Transmitted Infections (STIs) in Men Who Have Sex with Men and using oral TDF/FTC for HIV Pre-Exposure Prophylaxis (PrEP) and vaccination with Bexsero.

DETAILED DESCRIPTION:
This is a randomized study with a factorial design for the 2 biomedical interventions (interventions 1 and 2).

Subjects will be randomized and assigned to two different interventions:

* Intervention 1: PEP with doxycycline or no PEP. Subjects will be randomized 2/1 to receive doxycycline PEP or no PEP
* Intervention 2: Meningococcal B vaccine (Bexsero®) or no vaccine Subjects will be randomized 1/1 to received 2 doses of Bexsero® vaccine (at the first visit and two months later) or no vaccine

Participants will be randomized in one of the following arms:

* Arm 1: doxycycline and Bexsero® vaccine (240 participants)
* Arm 2: doxycycline and no Bexsero® vaccine (240 participants)
* Arm 3: no doxycycline and Bexsero® vaccine (120 participants)
* Arm 4: no doxycycline and no Bexsero® vaccine (120 participants)

Randomization will be stratified by whether or not the participant enters in the ancillary study "intestinal microbiota".

ELIGIBILITY:
Inclusion Criteria:

* Mens who have sex with mens (MSM) enrolled in the ANRS PREVENIR study.
* At least 6-month experience with PrEP (within the ANRS PREVENIR study or before starting the ANRS PREVENIR study).
* No clinical manifestation of primary HIV infection and no symptom of bacterial STI (chlamydia, gonorrhea, M. genitalium or syphilis).
* History of documented bacterial STI with at least one episode in the last 12 months.
* Participants who agree to sign the information and consent form specific to this study.
* Valid health insurance (State medical aid (AME) is not health insurance).

Exclusion Criteria:

* Syphilis diagnosed prior to inclusion without serologic evidence of cure (cure is defined as decreased by at least 4-fold of the non-treponemal antibody titer [Venereal Disease Research Laboratory (VDRL), Rapid Plasma Reagin (RPR)] relative to the titer at initiation of treatment of syphilis).
* HIV infection.
* Previous vaccination with Bexsero® or any other meningococcal B vaccine.
* Vaccination during the 4 weeks (28 days) preceding the first vaccination of the study.
* Previous vaccination with an experimental vaccine in the previous 5 years.
* Systemic treatment with retinoids : isotretinoin (Acnetrait®, Procuta®, Curacné®, Contracné®, …).
* Treatment with enzyme-inducing anticonvulsants (carbamazepine, phenobarbital, phenytoin, ….).
* Participant who has received immunoglobulins, a transfusion of blood or blood derivatives in the last 3 months.
* Known or suspected congenital or acquired immunodeficiency; immunosuppressive treatment in the last 6 months, such as cancer chemotherapy or radiotherapy; long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks in the last 3 months)
* Known allergy to antibiotics of the tetracycline family.
* Known allergy to any component of the Bexsero® vaccine.
* Known allergy to any component of the doxycycline pill.
* Known allergy to latex (contained in the vaccine cap).
* Thrombocytopenia or any other known coagulation disorder, which would be a contraindication to an intramuscular injection of Bexsero® vaccine.
* Documented oesophageal lesion
* Acute respiratory infection or severe acute febrile illness or systemic reaction that may present a significant risk if vaccinated in the month prior to inclusion.
* Any condition (clinical) that, in the investigator's opinion, would contraindicate intramuscular vaccination and blood sampling.
* Oral Anticoagulant treatment.
* Continuous treatment with doxycycline at inclusion.
* Vitamin A treatment in case of intake of 10 000 international unit or more.
* Participation in another research including an exclusion period still in progress at the time of inclusion.
* Under guardianship or curator, or deprived of liberty by a judicial or administrative decision.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-02-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
For intervention 1 (with or without doxycycline PEP) : 1st occurence of chlamydia or syphilis after the enrolment visit (Day 0) | Month 24
  Intervention 1 (with or without doxycycline PEP) is the first episode of chlamydia or syphilis after the enrolment visit (Day 0) (chlamydia and syphilis diagnosed at the enrolment visit will not be included in the primary endpoint).
  Chlamydia détection will be performed by polymerase chain reaction.Syphilis détection will be performed by antigen.
For intervention 2 with or without Bexsero® vaccine : 1st occurence of gonorrhea reported one month after the second vaccine injection | Month 24
  Intervention 2 (with or without Bexsero® vaccine) is the first episode of gonorrhea reported one month after the second vaccine injection, so starting at the month 3 visit (gonorrhea episodes diagnosed at the enrolment visit and before the month 3 visit will not be included in the primary endpoint).
  In these analyses, subject follow-up will be right-censored at the time of the first STI.
  Gonorrhea détection will be performed by polymerase chain reaction.

SECONDARY OUTCOMES:
- Occurrence of a first episode of each of the bacterial STIs as well as cumulative incidence of each bacterial STIs | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  - Occurrence of a first episode of each of the bacterial STIs as well as cumulative incidence of each bacterial STIs (syphilis, chlamydia; gonorrhoea and Mycoplasma genitalium) during the trial. In that case, the entire follow-up will be considered.
  Chlamydia détection will be performed by polymerase chain reaction. Syphilis détection will be performed by antigen.
  Mycoplasma genitalium be performed by polymerase chain reaction. Gonorrhea détection will be performed by polymerase chain reaction.
- Occurrence of a new episode of anal or urinary gonorrhoea. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  - Occurrence of a new episode of anal or urinary gonorrhoea. Gonorrhea détection will be performed by polymerase chain reaction.
- Occurrence of a first symptomatic episode of chlamydia infection or gonorrhea | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  - Occurrence of a first symptomatic episode of chlamydia infection or gonorrhea at urinary or anal sites.
  Chlamydia détection will be performed by polymerase chain reaction. Gonorrhea détection will be performed by polymerase chain reaction.
- Proportion of patient with Methicillin-Resistant Staphylococcus Aureus and/or doxycycline resistant Staphylococcus aureus from throat. Fecal carriage of Extended-Spectrum Beta-Lactamase-producing Enterobacteriaceae Composition of intestinal microbiota | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  detection from throat swab of carriage of MRSA (methicillin-resistant Staphylococcus aureus) and/or doxycycline resistant Staphylococcus aureus, fecal carriage of ESBL (extended-spectrum beta-lactamase) -producing Enterobacteriaceae, and composition of the intestinal microbiota), all détected by polymerase chain reaction assay
- Incidence of clinical and biological adverse events | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  Proportion of patients experiencing a clinical or biological adverse events (ANRS scale)
- Proportion of patients taking doxycycline | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  Adherence will be evaluated by doxycycline pills taken by patients
- Concentration of doxycycline in hair | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  Adherence will be evaluated by détection of doxycyclin in hair
- Proportion of patients with Antibiotic susceptibilities of all strains of NG (Neisseria gonorrhoeae), CT (chlamydiae trachomatis), MG (mycoplasma genitalium) | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  identification of Antibiotic susceptibilities of all strains of NG (Neisseria gonorrhoeae), CT (chlamydiae trachomatis), MG (mycoplasma genitalium) to doxycycline, macrolides, fluoroquinolones and third generation cephalosporin will be performed by PCR (polymerase chain reaction assay)
- Rate of cured STIs after treatment with or without PEP. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  declaration of illnesses from infection to healing
- Incidence of resistance to antibiotics of Neisseria gonorrhoeae with or without doxycycline. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  Proportion of participants with resistance to antibiotics of Neisseria gonorrhoeae will be evaluated by polymerase chain reaction to detect mutations
- Incidence of Serum bactericidal activity against meningococcal and gonococcal antigens over time in participants of Bexsero®'s arm. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  Proportion of participants with Serum bactericidal activity against meningococcal and gonococcal antigens
- Incidence of clinical and biological adverse events following Bexsero® vaccine. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  Proportion of participants experiencing a clinical and biological adverse events following Bexsero® vaccine (ANRS scale)
- Prevalence and incidence of meningococcal carriage in pharyngeal, anal and urine swabs. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  detection of meningococcal carriage in pharyngeal, anal and urine swabs will be performed
- Impact of PEP or Bexsero® vaccine on sexual behaviour | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  rates of condom use for receptive anal intercourse, number of sexual partners and number of sex acts over time
- Incidence of HIV infection with both prophylaxis strategies. | Month 2, Month 3, Month 6, Month 12, Month 18, Month 21, Month 24
  HIV infection will be tested by serology and western blot assay

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Hôpital Bichat, Paris
  - Hôpital Hôtel Dieu, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital pitié Salpetrière, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris

REFERENCES:
- [Derived] Molina JM, Bercot B, Assoumou L, Rubenstein E, Algarte-Genin M, Pialoux G, Katlama C, Surgers L, Bebear C, Dupin N, Ouattara M, Slama L, Pavie J, Duvivier C, Loze B, Goldwirt L, Gibowski S, Ollivier M, Ghosn J, Costagliola D; ANRS 174 DOXYVAC Study Group. Doxycycline prophylaxis and meningococcal group B vaccine to prevent bacterial sexually transmitted infections in France (ANRS 174 DOXYVAC): a multicentre, open-label, randomised trial with a 2 x 2 factorial design. Lancet Infect Dis. 2024 Oct;24(10):1093-1104. doi: 10.1016/S1473-3099(24)00236-6. Epub 2024 May 23. PMID 38797183